CLINICAL TRIAL: NCT01871506
Title: Integrating Tobacco Treatment Into Cancer Care: A Randomized Controlled Comparative Effectiveness Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Elyse Park, PhD, Associate Professor of Psychiatry, Harvard Medical School, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013P001036; 1R01CA166147-01A1 (NIH)
Record Dates: First submitted 2013-06-04; First posted 2013-06-06 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Care (SC) (Experimental): Participants randomized to "standard care" (SC) will have the option to receive 4 behavioral counseling sessions with a tobacco treatment counselor and medication advice.
  Interventions: Behavioral: Standard Care (SC)
- Intensive Counseling (IC) (Experimental): Participants randomized to intensive counseling (IC) will receive the same 4 initial behavioral counseling sessions with a tobacco treatment counselor as participants in the SC arm. IC participants have the option to also receive:
  * Extended Counseling: An additional 4 biweekly and 3 monthly proactive counseling sessions with a tobacco treatment counselor (total of 11 counseling contacts).
  * Smoking Cessation Medication: Up to a 12-week supply of FDA approved smoking cessation medication [varenicline, bupropion, or combination NRT (patch + lozenge)] at no cost to the participant.
  Interventions: Behavioral: Intensive Counseling (IC)

INTERVENTIONS:
Behavioral: Standard Care (SC) — 1. Initial counseling session: The initial counseling session will last approximately 45 minutes and will be conducted in-person or by phone by a tobacco treatment counselor. The session will be structured in a 5 As format and utilize Motivational Interviewing (MI) techniques.
  2. 3 Weekly Follow-up Counseling Sessions: SC Patients will be offered 3 weekly proactive follow-up sessions, concentrated on quitting and staying quit throughout cancer treatment.
  3. Medication advice: The tobacco counselor will advise SC subjects to use smoking cessation medication to assist with their quit. Smoking cessation medication will not be provided by the study free of cost for SC subjects.
  Other Names: "Standard of Care" Treatment
  Arms: Standard Care (SC)
Behavioral: Intensive Counseling (IC) — The IC model includes all components of the SC as well as extended counseling support and up to 90 days of free FDA approved smoking cessation medication.
  1. Extended counseling support: Participants in the IC group will be offered the same initial 4 counseling sessions as the SC group as well as 4 additional proactive biweekly sessions and 3 monthly booster sessions.
  2. Smoking cessation medication: IC participants will be offered a 4-week supply of FDA-approved smoking cessation medication (varenicline, bupropion or nicotine replacement therapy) of their choice, with the option to renew the medication twice for up to 90 days of free medication. Participants are not required to take smoking cessation medication.
  Other Names: Intensive Treatment
  Arms: Intensive Counseling (IC)

SUMMARY:
There are currently over 11 million cancer survivors in the U.S. and survival rates are increasing. Unfortunately, 10-30% of cancer patients are current smokers at the time of diagnosis, and many of these patients have elevated socioeconomic, medical, and psychosocial vulnerabilities. Documented risks associated with continued smoking following cancer diagnosis include decreased survival time; increased complications from surgery, radiation, and chemotherapy; and increased risk of second primary tumors. U.S. Department of Health & Human Services Public Health Service evidence-based tobacco treatment guidelines exist but have not been integrated into the cancer setting. This is a tremendous missed opportunity to address a modifiable risk factor. In recognition of this treatment gap, the National Cancer Institute (NCI) sponsored a conference in 2009 to address how to increase the readiness and capacity for delivery of tobacco treatment in Cancer Centers. The American Society of Clinical Oncology (ASCO) recommends identification, advice, and counseling of all smokers by their second oncology visit as a core quality indicator; however, currently only half of patients report being asked about tobacco use.

Specific Aim: To conduct a randomized controlled comparative effectiveness trial of two strategies to promote smoking cessation in suspected or newly diagnosed cancer patients.

Study Design: A multi-site randomized controlled comparative effectiveness trial will enroll 295 current smokers with suspected or newly diagnosed melanoma, lymphoma, thoracic, breast, genitourinary, gastrointestinal, head and neck, or gynecologic cancer. Participants will be randomly assigned to receive Intensive Counseling (IC) or "Standard Care" (SC). Both groups will receive an initial motivational counseling session and 3 weekly follow-up counseling sessions with a tobacco treatment counselor, conducted in-person or by telephone. The IC arm has the option to also receive:

* Smoking Cessation Medication: Up to a 12-week supply of FDA approved smoking cessation medication (Varenicline, bupropion, or combination NRT) at no cost to the participant.
* Extended Counseling: An additional 4 biweekly and 3 monthly proactive counseling sessions with a tobacco treatment counselor (total of 11 counseling contacts).

All participants will complete 1 baseline and 2 follow-up surveys, at 3 and 6 months. Self-reported abstinence will be biochemically confirmed at 3 and 6 months.

DETAILED DESCRIPTION:
Specific Aims

Aim 1: To compare the effectiveness of two tobacco treatments that are integrated into cancer care in producing tobacco abstinence at 6 months.

Aim 2: To explore: a) mechanisms through which treatment promotes abstinence; b) subpopulations in which abstinence is promoted; and c) which aspects of treatment promote abstinence.

Aim 3: To compare the incremental cost effectiveness (cost per quit) of two tobacco treatments.

Exploratory Aim: To identify the percentage and associated characteristics of smokers who 1) enroll in tobacco treatment and 2) adhere to tobacco treatment.

ELIGIBILITY:
INCLUSION CRITERIA:

Adult men and women may participate in this study if he/she meet the following requirements:

1. Current, new* patient at one of our three participating study sites: Massachusetts General Hospital (MGH) Cancer Center, Memorial Sloan Kettering Cancer Center (MSKCC), or Dana-Farber Cancer Institute (DFCI);
2. Currently with suspected or newly diagnosed cancer (thoracic, breast, genitourinary, gastrointestinal, head and neck, gynecologic, lymphoma, melanoma);
3. Has smoked a cigarette, even a puff, in the past 30 days;
4. Is willing to consider trying to quit smoking using counseling and/or smoking cessation medication;
5. Is English or Spanish speaking (MGH); English speaking (MSK; DFCI);
6. Has regular telephone access.

[*Patients will be considered "new" and eligible under the following conditions:

1. if they are attending approximately one of their first 4 visits or are within approximately 3 months of the initial visit date with their primary oncologist at the Massachusetts General Hospital (MGH) Cancer Center, Memorial Sloan Kettering Cancer Center (MSKCC), or Dana-Farber Cancer Institute (DFCI) for suspected or recently diagnosed cancer;
2. if they come to the MGH, MSKCC, or DFCI for a second opinion, the patient opts to receive their cancer treatment at any of these institutions;
3. if they have a past cancer diagnosis, they are currently faced with a local and distant recurrence of tumors;
4. if they have been treated previously for other types of cancer, they are currently faced with a new form of cancer.]

EXCLUSION CRITERIA:

In an effort to be as inclusive as possible, a patient will be excluded only if he/she:

1. Is NOT currently receiving or has no intentions to receive care at one of three participating cancer treatment centers: Massachusetts General Hospital Cancer Center, Memorial Sloan Kettering Cancer Center, or Dana-Farber Cancer Institute (DFCI);
2. Is currently psychiatrically unstable or otherwise unable to provide informed consent as determined by study investigators or oncology clinician;
3. Is not English or Spanish speaking;
4. Is medically ineligible (as determined by their treating physician);
5. Has insufficient comprehension/literacy.

ADDITIONAL INFORMATION:

Participant inclusion/exclusion is not based on use of smoking cessation medication -- he/she may decide not to use any smoking cessation medication and still participate in the study. Patients deemed ineligible will be referred to the state quit line.

Patients interested in participating in the study should contact the appropriate contact person, based on whether they are a current patient at the MGH, MSKCC, or DFCI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elyse R Park, Ph.D., MPH, Principal Investigator — Massachusetts General Hospital; Jamie S. Ostroff, Ph.D., Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Park ER, Perez GK, Regan S, Muzikansky A, Levy DE, Temel JS, Rigotti NA, Pirl WF, Irwin KE, Partridge AH, Cooley ME, Friedman ER, Rabin J, Ponzani C, Hyland KA, Holland S, Borderud S, Sprunck K, Kwon D, Peterson L, Miller-Sobel J, Gonzalez I, Whitlock CW, Malloy L, de Leon-Sanchez S, O'Brien M, Ostroff JS. Effect of Sustained Smoking Cessation Counseling and Provision of Medication vs Shorter-term Counseling and Medication Advice on Smoking Abstinence in Patients Recently Diagnosed With Cancer: A Randomized Clinical Trial. JAMA. 2020 Oct 13;324(14):1406-1418. doi: 10.1001/jama.2020.14581. PMID 33048154
- [Derived] Park ER, Ostroff JS, Perez GK, Hyland KA, Rigotti NA, Borderud S, Regan S, Muzikansky A, Friedman ER, Levy DE, Holland S, Eusebio J, Peterson L, Rabin J, Miller-Sobel J, Gonzalez I, Malloy L, O'Brien M, de Leon-Sanchez S, Whitlock CW. Integrating tobacco treatment into cancer care: Study protocol for a randomized controlled comparative effectiveness trial. Contemp Clin Trials. 2016 Sep;50:54-65. doi: 10.1016/j.cct.2016.07.016. Epub 2016 Jul 19. PMID 27444428

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 11/25/2013 and 7/1/2017 4709 patients were screened for eligibility. 2659 were eligible based on screen criteria; 1808 did not complete the screen. Of the 851 who were approached to complete the screen, 405 were ineligible, 303 enrolled and were randomized, and 143 refused (84 refused consent and 59 did not complete the baseline survey)
Pre-assignment Details: Of the 446 eligible for the study, 303 were randomized, 84 were eligible but refused consent (top 3 reasons: too upset, did not need help, had no time) and 59 were eligible but were not randomized because they did not complete a baseline survey.
Groups:
- Standard Treatment (ST): Participants randomized to "standard treatment" will have the option to receive 4 behavioral counseling sessions with a tobacco treatment counselor and medication advice.
  Standard Treatment (ST): (1) Initial counseling session: The initial counseling session will last approximately 45 minutes and will be conducted in-person or by phone by a tobacco treatment counselor. The session will be structured in a 5 As format and utilize Motivational Interviewing (MI) techniques.
  (2) 3 Weekly Follow-up Counseling Sessions: SC Patients will be offered 3 weekly proactive follow-up sessions, concentrated on quitting and staying quit throughout cancer treatment.
  (3) Medication advice: The tobacco counselor will advise SC subjects to use smoking cessation medication to assist with their quit. Smoking cessation medication will not be provided by the study free of cost for SC subjects.
- Intensive Treatment (IT): Participants randomized to intensive treatment (IT) will receive the same 4 initial behavioral counseling sessions with a tobacco treatment counselor as participants in the ST arm. IT participants have the option to also receive:
  * Extended Counseling: An additional 4 biweekly and 3 monthly proactive counseling sessions with a tobacco treatment counselor (total of 11 counseling contacts).
  * Smoking Cessation Medication: Up to a 12-week supply of FDA approved smoking cessation medication [varenicline, bupropion, or combination NRT (patch + lozenge)] at no cost to the participant.
  Intensive Treatment (IT): The IT model includes all components of the ST as well as extended counseling support and up to 90 days of free FDA approved smoking cessation medication.
Period: Overall Study
Arm/Group | Standard Treatment (ST) | Intensive Treatment (IT)
Started | 150 | 153
Completed | 150 | 153
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Standard Treatment (ST): Participants randomized to "standard treatment" will have the option to receive 4 behavioral counseling sessions with a tobacco treatment counselor and medication advice.
  Standard Treatment (ST): (1) Initial counseling session: The initial counseling session will last approximately 45 minutes and will be conducted in-person or by phone by a tobacco treatment counselor. The session will be structured in a 5 As format and utilize Motivational Interviewing (MI) techniques.
  (2) 3 Weekly Follow-up Counseling Sessions: ST Patients will be offered 3 weekly proactive follow-up sessions, concentrated on quitting and staying quit throughout cancer treatment.
  (3) Medication advice: The tobacco counselor will advise SC subjects to use smoking cessation medication to assist with their quit. Smoking cessation medication will not be provided by the study free of cost for SC subjects.
- Intensive Treatment (IT): Participants randomized to intensive treatment (IT) will receive the same 4 initial behavioral counseling sessions with a tobacco treatment counselor as participants in the SC arm. IC participants have the option to also receive:
  * Extended Counseling: An additional 4 biweekly and 3 monthly proactive counseling sessions with a tobacco treatment counselor (total of 11 counseling contacts).
  * Smoking Cessation Medication: Up to a 12-week supply of FDA approved smoking cessation medication [varenicline, bupropion, or combination NRT (patch + lozenge)] at no cost to the participant.
  Intensive Counseling: The IT model includes all components of the ST as well as extended counseling support and up to 90 days of free FDA approved smoking cessation medication.
- Total: Total of all reporting groups
Arm/Group | Standard Treatment (ST) | Intensive Treatment (IT) | Total
Number analyzed (Participants) | 150 | 153 | 303
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (9.5) | 58 (9.9) | 58 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 87 | 170
  Male | 67 | 66 | 133
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 7 | 11
  Not Hispanic or Latino | 146 | 146 | 292
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 17 | 14 | 31
  White | 131 | 134 | 265
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 150 | 153 | 303

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Biochemically Verified 7-day Point Prevalence Tobacco Abstinence at 6 Months
Description: Number of participants with 7-day point-prevalence tobacco abstinence at 6-month follow-up, assessed by biochemically confirmed saliva cotinine (<15 ng/ml76, 82) or <10 ppm expired air carbon monoxide (CO) for participants concurrently using NRT
Time Frame: 6 months
Population: Twenty participants were too ill or deceased to complete follow-up assessment. Given the study participant population of cancer patients, our trial was powered accounting for cancer deaths and reporting participants who were alive at follow-up assessment.
Measure: Count of Participants; unit: Participants
Groups:
- Standard Treatment (ST): Participants randomized to "standard treatment" (ST) will have the option to receive 4 behavioral counseling sessions with a tobacco treatment counselor and medication advice.
  Standard Treatment (ST): (1) Initial counseling session: The initial counseling session will last approximately 45 minutes and will be conducted in-person or by phone by a tobacco treatment counselor. The session will be structured in a 5 As format and utilize Motivational Interviewing (MI) techniques.
  (2) 3 Weekly Follow-up Counseling Sessions: SC Patients will be offered 3 weekly proactive follow-up sessions, concentrated on quitting and staying quit throughout cancer treatment.
  (3) Medication advice: The tobacco counselor will advise SC subjects to use smoking cessation medication to assist with their quit. Smoking cessation medication will not be provided by the study free of cost for SC subjects.
- Intensive Treatment (IT): Participants randomized to the Intensive Treatment (IT) will receive the same 4 initial behavioral counseling sessions with a tobacco treatment counselor as participants in the SC arm. IT participants have the option to also receive:
  * Extended Counseling: An additional 4 biweekly and 3 monthly proactive counseling sessions with a tobacco treatment counselor (total of 11 counseling contacts).
  * Smoking Cessation Medication: Up to a 12-week supply of FDA approved smoking cessation medication [varenicline, bupropion, or combination NRT (patch + lozenge)] at no cost to the participant.
  Intensive Counseling (IC): The IC model includes all components of the SC as well as extended counseling support and up to 90 days of free FDA approved smoking cessation medication.
  (1) Extended counseling support: Participants in the IC group will be offered the same initial 4 counseling sessions as the SC group as well as 4 additional proactive biweekly sessions and 3 monthly booster sessions.
Arm/Group | Standard Treatment (ST) | Intensive Treatment (IT)
Number analyzed (Participants) | 135 | 148
Participants | 29 | 51

2. Secondary Outcome: Number of Participants With Biochemically Verified 7-day Point Prevalence Tobacco Abstinence at 3 Months
Description: Number of participants with7 -day point-prevalence tobacco abstinence at 3-month follow-up, assessed by biochemically confirmed saliva cotinine (<15 ng/ml76, 82) or <10 ppm expired air carbon monoxide (CO) for participants concurrently using NRT
Time Frame: 3 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Standard Treatment (ST): Participants randomized to ST will have the option to receive 4 behavioral counseling sessions with a tobacco treatment counselor and medication advice.
  Standard Care (SC): (1) Initial counseling session: The initial counseling session will last approximately 45 minutes and will be conducted in-person or by phone by a tobacco treatment counselor. The session will be structured in a 5 As format and utilize Motivational Interviewing (MI) techniques.
  (2) 3 Weekly Follow-up Counseling Sessions: SC Patients will be offered 3 weekly proactive follow-up sessions, concentrated on quitting and staying quit throughout cancer treatment.
  (3) Medication advice: The tobacco counselor will advise SC subjects to use smoking cessation medication to assist with their quit. Smoking cessation medication will not be provided by the study free of cost for SC subjects.
- Intensive Treatment (IT): Participants randomized to IT will receive the same 4 initial behavioral counseling sessions with a tobacco treatment counselor as participants in the SC arm. IC participants have the option to also receive:
  * Extended Counseling: An additional 4 biweekly and 3 monthly proactive counseling sessions with a tobacco treatment counselor (total of 11 counseling contacts).
  * Smoking Cessation Medication: Up to a 12-week supply of FDA approved smoking cessation medication [varenicline, bupropion, or combination NRT (patch + lozenge)] at no cost to the participant.
Arm/Group | Standard Treatment (ST) | Intensive Treatment (IT)
Number analyzed (Participants) | 135 | 148
Participants | 28 | 46

3. Secondary Outcome: Number of Participants With Continuous Tobacco Abstinence
Description: Number of Participants with Continuous tobacco abstinence (between quit and follow-up) at 3 & 6 months
Time Frame: 3 months to 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Standard Treatment: Participants randomized to ST will have the option to receive 4 behavioral counseling sessions with a tobacco treatment counselor and medication advice.
  .
- Intensive Treatment): Participants randomized to intensive counseling IT will receive the same 4 initial behavioral counseling sessions with a tobacco treatment counselor as participants in the ST ar,m.
Arm/Group | Standard Treatment | Intensive Treatment)
Number analyzed (Participants) | 135 | 148
Participants | 26 | 43

4. Secondary Outcome: Number of Participants With Sustained Tobacco Abstinence
Description: Number of Participants with Biochemically confirmed repeated point prevalence abstinence at 3 & 6 months
Time Frame: 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Standard Treatment (ST): Participants randomized to ST will have the option to receive 4 behavioral counseling sessions with a tobacco treatment counselor and medication advice.
  .
- Intensive Treatment (IT): Participants randomized to IT will receive the same 4 initial behavioral counseling sessions with a tobacco treatment counselor as participants in the SC arm. IC participants have the option to also receive:
  .
Arm/Group | Standard Treatment (ST) | Intensive Treatment (IT)
Number analyzed (Participants) | 135 | 148
Participants | 17 | 35

5. Secondary Outcome: Number of Participants With Self-reported 7-day Point Prevalence.
Description: Number of Participants with Self-reported smoking abstinence of at least 7 days
Time Frame: 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Intensive Treatment (IT): Participants randomized to IT will receive the same 4 initial behavioral counseling sessions with a tobacco treatment counselor as participants in the SC arm. IC participants have the option to also receive:
Arm/Group | Standard Treatment (ST) | Intensive Treatment (IT)
Number analyzed (Participants) | 135 | 148
Participants | 42 | 54

6. Secondary Outcome: The Number of IT Participants Who Used Smoking Cessation Pharmacotherapy
Description: The number of IT participants who used 1) smoking cessation pharmacotherapy (Y/N dispensed) 2) smoking cessation counseling (Y/N), 3) 1-2 4-week refills, 4) took 1-3 monthly booster sessions.
Time Frame: Treatment Initiation to 6 month follow-up
Population: Only assessed intensive treatment arm.
Measure: Count of Participants; unit: Participants
Groups:
- Standard Treatment (ST): Participants randomized to ST will have the option to receive 4 behavioral counseling sessions with a tobacco treatment counselor and medication advice.
  S.
Arm/Group | Standard Treatment (ST) | Intensive Treatment (IT)
Number analyzed (Participants) | 0 | 153
Participants |  | 122

7. Secondary Outcome: The Number of IT Participants Who Used Smoking Cessation Counseling
Description: The number of intervention participants who used smoking cessation counseling during the study (Y/N)
Time Frame: Treatment Initiation to 6 Month Follow-up
Population: Only assessed intensive treatment arm
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Treatment (ST) | Intensive Treatment (IT)
Number analyzed (Participants) | 0 | 153
Participants |  | 153

8. Secondary Outcome: The Number of IT Participants Who Took 1-2 4-week Refills
Description: The number of intervention participants who took 1-2 4-week refills of smoking cessation medication
Time Frame: Treatment Initiation to 6 Month Follow-up
Population: Only assessed intensive treatment arm
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Treatment (ST) | Intensive Treatment (IT)
Number analyzed (Participants) | 0 | 153
Participants |  | 87

9. Secondary Outcome: The Number of IT Participants Who Took 1-3 Monthly Booster Sessions
Description: The number of IT participants who took 1-3 monthly booster sessions of smoking cessation counseling
Time Frame: Treatment Initiation to 6 Month Follow-up
Population: Only assessed intensive treatment arm
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Treatment (ST) | Intensive Treatment (IT)
Number analyzed (Participants) | 0 | 153
Participants |  | 99

10. Secondary Outcome: Cost-effectiveness
Description: The cost of the standard of care treatment and the cost of the intensive treatment.
Time Frame: 6 months
Population: Cost per quit (in dollars) are shown below.
Measure: Mean (95% Confidence Interval); unit: dollars
Groups:
- Intensive Treatment: Participants randomized to IT will receive the same 4 initial behavioral counseling sessions with a tobacco treatment counselor as participants in the SC arm. IC participants have the option to also receive:
  .
Arm/Group | Standard Treatment (ST) | Intensive Treatment
Number analyzed (Participants) | 150 | 153
dollars | 638 [570 to 710] | 1144 [1061 to 1231]

ADVERSE EVENTS:
Time Frame: Adverse events for each participant was collected over a 6-month period: from baseline to 6 month follow-up.
Description: Adverse events: Any untoward or unfavorable medical occurrence in a human subject including any abnormal sign, symptom, or disease...whether or not associated with the subject's participation in research. *Adverse events that are expected (i.e., documented in the protocol) are not reported to the IRB. More than one adverse event could be reported per participant.
Groups:
- Intensive Treatment (IT): Participants randomized to intensive treatment (IT) will receive the same 4 initial behavioral counseling sessions with a tobacco treatment counselor as participants in the SC arm. IT participants have the option to also receive:
  * Extended Counseling: An additional 4 biweekly and 3 monthly proactive counseling sessions with a tobacco treatment counselor (total of 11 counseling contacts).
  * Smoking Cessation Medication: Up to a 12-week supply of FDA approved smoking cessation medication [varenicline, bupropion, or combination NRT (patch + lozenge)] at no cost to the participant.
  I
Arm/Group | Standard Treatment (ST) | Intensive Treatment (IT)
All-Cause Mortality (participants affected / at risk) | 9/150 | 4/153
Serious Adverse Events (participants affected / at risk) | 0/150 | 0/153
Other Adverse Events (participants affected / at risk) | 17/150 | 41/153
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Treatment (ST) (N=150) | Intensive Treatment (IT) (N=153)
Nausea (General disorders) | 6 (6) | 13 (13) — General nausea, nausea and upset stomach, nausea and vomiting, nausea and increased heart rate related to smoking cessation medication use
Rash (General disorders) | 1 (1) | 4 (4) — Rash related to smoking cessation medication
Hiccups (General disorders) | 1 (1) | 3 (3) — Hiccups related to use of smoking cessation medication
SIADH (General disorders) | 0 (0) | 2 (2) — SIADH reaction to smoking cessation medication use
Bad taste in mouth (General disorders) | 0 (0) | 1 (1) — Bad taste in mouth related to smoking cessation medication
Flatulence (General disorders) | 1 (1) | 1 (1) — Flatulence related to smoking cessation medication
Mouth irritation (General disorders) | 0 (0) | 4 (4) — Mouth irritation, burning sensation in mouth, tingling sensation on tongue related to smoking cessation medication
Difficulty sleeping (General disorders) | 2 (2) | 3 (3) — Difficulty sleeping related to smoking cessation medication
Fatigue (General disorders) | 0 (0) | 1 (1) — Fatigue or fog-headedness related to smoking cessation medication
Chest discomfort (General disorders) | 0 (0) | 1 (1) — Chest discomfort or palpitations related to smoking cessation medication
Pain in lower back and leg (General disorders) | 0 (0) | 1 (1) — Pain in lower back and leg related to smoking cessation medication
Headache (General disorders) | 2 (2) | 1 (1) — Headache and headache with diarrhea related to smoking cessation medication
Heartburn (General disorders) | 1 (1) | 0 (0) — Heartburn related to smoking cessation medication
Lightheadedness (General disorders) | 0 (0) | 1 (1) — Lightheadedness related to smoking cessation medication
Swollen ankles (General disorders) | 1 (1) | 0 (0) — Swollen ankles related to smoking cessation medication
Vivid dreams (General disorders) | 2 (2) | 3 (3) — Vivid dreams related to smoking cessation medication
Malaise (General disorders) | 0 (0) | 1 (1) — Malaise related to smoking cessation medication
Shortness of breath (General disorders) | 0 (0) | 1 (1) — Shortness of breath related to smoking cessation medication

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-10): https://cdn.clinicaltrials.gov/large-docs/06/NCT01871506/Prot_SAP_000.pdf